CLINICAL TRIAL: NCT04932889
Title: Musculoskeletal Symptoms and Related Factors in Post Acute Covid-19 Patients
Brief Title: Musculoskeletal Symptoms in Post Acute Covid-19 Patients
Status: Completed | Type: Observational
Sponsor: Eskisehir City Hospital (Other)
Responsible Party: Principal Investigator, Fulya Bakılan, Specialist in physical medicine and rehabilitation, Eskisehir City Hospital
Other Study IDs: EskisehirCityH
Record Dates: First submitted 2021-06-14; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Covid19; Musculoskeletal Abnormalities
MeSH Terms: conditions — COVID-19; Musculoskeletal Abnormalities | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Change: the patients whose musculoskeletal symptoms initiated or aggravated with Covid-19 (n=240)
  Interventions: Other: Survey; Other: Laboratory parameters; Other: chest computed tomography
- No change: the patients whose musculoskeletal symptoms did not change with Covid-19 (n=40)
  Interventions: Other: Survey; Other: Laboratory parameters; Other: chest computed tomography

INTERVENTIONS:
Other: Survey — A detailed anamnesis was retrospectively recorded about age, gender, body mass index, education, working, the presence of any chronic disease (diabetes mellitus, hypertension, chronic obstructive pulmonary disease, cardiac disease, cancer, rheumatological disease…), smoking, duration of symptoms, usage of supplementing vitamins such as vitamin D,C, zinc…, treatment place (home quarantine, hospital, intensive care unit), duration of home quarantine and hospital treatment, the number of months since the onset of Covid-19 symptoms, usage of anticoagulants, treatment drugs such as hydroxychloroquine, favipiravir. Also the symptoms during the period of Covid-19 infection were recorded from patient files; cough, fever, dyspnea, chest pain, loss of smell and taste, sore throat, headache, no symptom, musculoskeletal symptoms such as: muscle, low back, back, joint pain.
Other: Laboratory parameters — The laboratory values of 182 patients, presence of chest computed tomography findings of 206 patients and symptoms of all patients during the period of Covid-19 infection, were retrospectively recorded. Laboratory values of hemoglobin, leucocyte, lymphocyte, platelet, C-reactive protein, erythrocyte sedimentation rate, ferritin, d-dimer, were recorded.
Other: chest computed tomography — Typical findings of chest CT were; bilateral, multifocal, peripheral ground glass opacities with/without consolidation, including the fissures, close to visceral pleural surfaces. Covid-19 Reporting and Data System (CO-RADS) was used for chest CT. CO-RADS assigns scores from 1 (very low suspicion of Covid-19) to 5 (very high suspicion of Covid-19).

SUMMARY:
The patients whose musculoskeletal symptoms initiated or aggravated with Covid-19, were compared with the patients whose musculoskeletal symptoms did not change with Covid-19. The variables; the demographic and treatment datas, admission symptoms, post acute-Covid-19 symptoms, laboratory, chest computed tomography findings.

DETAILED DESCRIPTION:
There is a lack of an overview of the factors associated with post acute-Covid-19 musculoskeletal symptoms. The aims are;1-to evaluate the most frequent admission symptoms and the frequency of musculoskeletal symptoms in post acute-Covid-19 patients,2-to determine the related factors with the post acute-Covid-19 musculoskeletal symptoms.

In this retrospective study; the patients whose musculoskeletal symptoms initiated or aggravated with Covid-19, were compared wthe patients whose musculoskeletal symptoms did not change with Covid-19. The variables; the demographic and treatment datas, admission symptoms, post acute-Covid-19 symptoms, laboratory (complete blood count, C-reactive protein, ferritin, D-dimer), chest computed tomography findings.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Having Covid-19 treatment (home quarantine / hospital / intensive care unit) according to a positive polymerase chain reaction (PCR) test in a nasopharyngeal + oropharyngeal swab or chest CT.

Exclusion Criteria:

* Patients who did not have musculoskeletal symptom records (admission symptoms and musculoskeletal symptoms such as; fatigue, spine / joint /muscle pain/ numbness) in patients files
* Acute Covid-19 patients whose symptoms started less than 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective cross-sectional study was carried out with the records of 280 post Covid-19 patients who admitted to the physical medicine and rehabilitation outpatient clinic between December 2020 and May 2021.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Rate of back pain | Baseline
  given as percentage %
Chest computed tomography | Baseline
  Presence of covid-19 findings in chest computed tomography (covid findings positive or negative)
Rate of low-back pain | Baseline
  given as percentage %
Rate of fatigue | Baseline
  given as percentage %
Rate of neck pain | Baseline
  given as percentage %
Rate of dyspnea | baseline
  given as percentage %
Rate of joint pain | Baseline
  given as percentage %
Rate of chest pain | Baseline
  given as percentage %
Rate of myalgia | Baseline
  given as percentage %

SECONDARY OUTCOMES:
age | Baseline
  years
Weight | Baseline
  kilograms
gender | Baseline
  female or male
Duration after the onset of covid-19 | Baseline
  months
Lymhocyte levels | Baseline
  10*3 cells/microliter
D-dimer levels | Baseline
  miligram/Litre
C-reactive protein | Baseline
  miligram/Litre
Hemoglobin | Baseline
  gram/desilitre
Platelet | Baseline
  10*3 cells/microliter
Ferritin | Baseline
  nanogram/mililitre

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Bakılan, Principal Investigator — Eskişehir City Hospital
Locations (1):
- Eskişehir City Hospital, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
one year later, after my manuscript publishes in a journal.